CLINICAL TRIAL: NCT01893957
Title: Evaluation of the Effects of High Voltage Electrical Stimulation in the Floe Blood and Tactile Sensitivity of Women Undergoing Axillary Lymphadenectomy
Brief Title: Effects of Electrical Stimulation on Blood Circulation and Sensibility Tactil in Lymphadenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, PhD, Professor, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1143-1024
Record Dates: First submitted 2013-06-21; First posted 2013-07-09 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; physical therapy; electrical stimulation; tactile sensitivity; flow blood
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy (Experimental): Healthy women undergoing high voltage electrical stimulation
  Interventions: Procedure: High voltage electrical stimulation - ( healthy women ); Device: Neurodyn High Volt Model (IBRAMED)
- Axillary lymphadenectomy (Experimental): Axillary lymphadenectomy volunteers undergoing to high voltage electrical stimulation
  Interventions: Procedure: high voltage electrical stimulation - axillary lymphadenectomy; Device: Neurodyn High Volt Model (IBRAMED)

INTERVENTIONS:
Procedure: high voltage electrical stimulation - axillary lymphadenectomy — Will be used high voltage electrical stimulation, Neurodyn High Volt Model (IBRAMED), twice a week, over the course of seven weeks,in 20-minute sessions on alternate days. The parameters are: high voltage pulsed current, monopolar (cathode), 100 Hz, synchronized mode, on/off relationship of 3:9 seconds, rise/decay 2:1 seconds, and motor threshold. The electrodes are positioned in the middle and distal thirds of the anterior surface of the forearm and arm.
  Arms: Axillary lymphadenectomy
Procedure: High voltage electrical stimulation - ( healthy women ) — Will be used high voltage electrical stimulation, Neurodyn High Volt Model (IBRAMED), twice a week, over the course of seven weeks,in 20-minute sessions on alternate days. The parameters are: high voltage pulsed current, monopolar (cathode), 100 Hz, synchronized mode, on/off relationship of 3:9 seconds, rise/decay 2:1 seconds, and motor threshold. The electrodes are positioned in the middle and distal thirds of the anterior surface of the forearm and arm.
  Arms: Healthy
Device: Neurodyn High Volt Model (IBRAMED)

SUMMARY:
The aim of this study is to investigate the influence of electrical stimulation at the speed of blood circulation and tactile sensitivity of the arms of women who underwent axillary dissection for breast cancer.

DETAILED DESCRIPTION:
Introduction: the surgical treatment of breast cancer, especially axillary lymphadenectomy (AL), can cause blood circulatory changes, also partial or total lesion of the sensory nerve intercostobrachial, often causing anesthesia or hypoesthesia in the corresponding dermatome ipsilateral upper limb surgery. Objective: to investigate the influence of high voltage electrical stimulation (HVES) in the in the blood flow and tactile sensitivity in nerve path intercostobrachial of women undergoing AL. Methodology: sample of 30 volunteers, aged between 40 and 60 years, divided into two equal groups (n = 15): women with axillary dissection for breast cancer undergoing therapeutic procedure (GAL) and control group (CG) composed of women who did not undergoing axillary surgery. The treatment procedure consist of the application of high voltage electrical simulation for 30 minutes in both limbs twice a week over the course of seven weeks. The profile of blood flow, including speed, direction were evaluated by means of continuous wave Doppler ultrasound. The assessment of tactile sensitivity was accomplished through esthesiometer in three stages: before the start of the first therapeutic procedure, after completion of the intervention and 30 days after the end of treatment (wash-out). The data will be analyzed using descriptive statistics (ANOVA) even as the hypothesis testing of Shapiro-Wilk and if the data are not normally distributed, non-parametric tests will be used. For the analyses will be used SPSS software with critical level of 5%. The results obtained on this study aim to justify therapies for intervention with that equipment in the treatment of morbidities caused by axillary linfadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* women, 40 to 60 years old, with abnormal sensitivity of the ipsilateral upper limb due to Type Madden Modified Radical Mastectomy for breast cancer with axillary lymphadenectomy

Exclusion Criteria:

* patients undergoing other types of surgery that is not considered in the inclusion criteria, bilateral mastectomy, has a diagnosis of metastases, and skin disorders such as ulcers or erysipelas in the region (or nearby) the intercostal nerve pathway. We also excluded volunteers with some sort of cognitive impairment

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Tactile sensitivity | 2 years
  Will be used Estesiômetro Semmes-Weinstein (SORRY®) to evaluate the tactile sensibility in dermatomes corresponding on the medial and superior-posterior arm.

SECONDARY OUTCOMES:
Blood flow velocity | 2 years
  The evaluation of the peripheral arterial and venous flow in the upper limbs will be accomplished through the equipment ultrasound Doppler (Nicolet Vascular Versalab SE®), and the collection site will be in the antecubital fossa, of the brachial artery and brachial vein.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil